CLINICAL TRIAL: NCT00643370
Title: Quantifying Lung Tumor Movement Under Dep Inspiration Breath Holds
Brief Title: Quantifying Lung Tumor Movement Under Deep Inspiration Breath Holds
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LU-23980
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2011-08

CONDITIONS: Lung Cancer
Keywords: lung cancer; tumor motion
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1: single arm study
  Interventions: Other: CT scan of the chest under deep inspiration breath hold

INTERVENTIONS:
Other: CT scan of the chest under deep inspiration breath hold — computed tomography scan of the chest under dep inspiration breath hold conditions

SUMMARY:
Radiotherapy is a common treatment for lung cancer. One Challenge of delivering radiation treatment to lung tumors accurately is tumor movement which occurs as a patient breathes. In some situations, tumors move enough during breathing so that some or all of the tumor may be missed by a radiation treatment. One way to decrease the amount a lung tumor moves during radiotherapy treatments is for patients to held their breath briefly during a radiation treatment. By doing this, a patient's lung tumor may not move as much as it would during regular breathing. In this study, the investigators aim to study patients with lung cancers which move during breathing. Patients will be asked to hold their breath after inspiration while a CT scan of their lung tumor is obtained. The purpose of this study is to study how much less patients' lung tumors move when they hold their breath

ELIGIBILITY:
Inclusion Criteria:

* biopsy confirmed primary lung cancer
* undergoing radiotherapy or chemoradiotherapy
* able to perform adequate deep inspiration breath hold
* patients of childbearing potential must practice adequate contraception
* signed study-specific informed consent form

Exclusion Criteria:

* unable to perform adequate deep inspiration breath hold
* prior tumor resection
* prior chest or neck RT
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with any primary lung cancer who are undergoing radiotherapy or chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
tumor movement | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, FRCPC, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada